CLINICAL TRIAL: NCT00135434
Title: Effect of HIV Protease Inhibitor Drugs on Glucose and Insulin Metabolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AI424-130
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2009-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; lopinavir-ritonavir drug combination

INTERVENTIONS:
Drug: Atazanavir/Ritonavir/Lopinavir/ritonavir

SUMMARY:
This study examined the effects of two commonly prescribed HIV drugs on the way the body metabolizes glucose, insulin and fat.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity by euglycemic hyperinsulinemic clamp method

SECONDARY OUTCOMES:
Insulin sensitivity by oral glucose tolerance
Lipids and lipoproteins

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Clinical Pharmacology Unit, Bristol-Myers Squibb Company, Hamilton, New Jersey, United States